CLINICAL TRIAL: NCT00743834
Title: Cost-Effectiveness of Adding Web-Based CBT to Luvox CR for OCD
Brief Title: Cost-Effectiveness of Adding Web-Based Cognitive-Behavioral Therapy (CBT) to Luvox CR for Obsessive Compulsive Disorder (OCD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rogers Center for Research & Training, Inc. (Other)
Responsible Party: John H Greist, MD, Rogers Center for Research & Training, Inc.
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: JIIT-07-LCR001a
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fluvoxamine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Effectiveness of Luvox CR plus Web-based CBT for OCD
  Interventions: Drug: Luvox CR; Behavioral: Behavioral Therapy

INTERVENTIONS:
Drug: Luvox CR — In light of the Luvox-CR dosing procedure of Hollander et al (2003) (50 mg increments weekly) and the available dose capsules of Luvox-CR (100 mg and 150 mg), the Luvox-CR dose will be increased over the first 6 weeks of treatment as tolerated in 50 mg to 100-mg increments every week, as tolerated and clinically indicated, to a bedtime dose between 100 and 300 mg/day. The dose will then be held constant for the duration of the study
Behavioral: Behavioral Therapy — The web-based CBT (CT STEPS) includes an introductory session explaining the treatment, with videotapes of OCD patients who used an earlier version, along with 9 subsequent treatment modules. The CBT will include weekly email feedback from a psychologist in response to questions asked about the CBT by the subjects assigned to this treatment arm.

SUMMARY:
This study will test the hypotheses that: 1. 12 weeks of Luvox-CR plus web-based Cognitive-Behavioral Therapy (CBT) [CT-STEPS] will produce greater symptom relief of OCD than treatment with Luvox-CR alone; and, 2. subjects receiving 12 weeks of CT-STEPS added to Luvox-CR treatment after 12-weeks of Luvox-CR monotherapy will experience greater OCD symptom relief (from weeks 12-24) than those continuing Luvox-CR treatment and having access to CT-STEPS from week one. 3. subjects who begin CT-STEPS at week 12 will be more likely to complete it than those who begin CT-STEPS at baseline.

DETAILED DESCRIPTION:
Primary Endpoint(s): Change in Y-BOCS score from baseline to endpoint at weeks 12 and 24; and, number (and percent) "responders" at weeks 12 and 24, defined as subjects with a 35% decrease in Y-BOCS score at endpoint and a Clinical Global Impressions score of 1 or 2 (very much or much improved).

Secondary Endpoint(s):

1. change in scores on the Work and Social Adjustment Scale, a quality of life measure
2. change in scores on the Work Productivity and Activity Impairment

   Questionnaire:

   Specific Health Problem scale; in particular, we will analyze change in work hours/week lost because of OCD, and change in effect of OCD on work productivity (0-10 scale).
3. dollar cost per responder
4. dollar cost per total number of patients needed to produce one additional responder in the Luvox-CR plus web-based CBT group over the number produced by Luvox-CR alone, i.e., dollar cost per number needed to treat
5. dollar cost per 5% decrease in Y-BOCS score at weeks 12 and 24 in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years, with OCD of at least 1 year's duration, meeting DSM-IV diagnostic criteria, and having a baseline Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score of 18.

Exclusion Criteria:

* Pregnant or nursing women or women of childbearing age not using an effective contraceptive method
* Organic mental disorder
* Bipolar disorder
* Psychotic disorder
* History of substance abuse or dependence within 3 years of evaluation for study
* Major depression with suicidal risk
* Major depression dominating the clinical picture
* Panic disorder
* Personality disorder severe enough to interfere with cooperation with study procedures
* Need for antipsychotic medication
* Depot neuroleptic drug within 6 months
* Fluoxetine within 5 weeks
* An MAOI within 2 weeks, any nightly sedative, or taking a medication that may interact with fluvoxamine
* Serious or unstable medical condition (hematological, endocrine, cardiovascular, renal or gastrointestinal), a history of malignancy (other than excised basal cell carcinoma), history of brain disease, including more than one childhood febrile convulsion and all forms of epilepsy; or, are receiving behavior therapy for OCD.
* Subjects who qualify for the study while taking an SSRI must have been taking their current dose or a higher dose for at least 12 weeks prior to study baseline.
* Subjects who qualify for the study while taking fluvoxamine must be taking no more than 150 mg/day and never had a trial at a higher dose, must be believed by the investigator to be able to tolerate an increase to 250 mg/day starting at baseline, and must have been taking their pre-study dose or a higher dose (up to 150 mg/day) for at least 12 weeks prior to study baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure (Y-BOCS score) will be obtained by clinician rating | screening, baseline, and end of weeks 4, 8, 12, 16, 20 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: John H Greist, MD, Principal Investigator — The Rogers Center for Research & Training, Inc.
Locations (1):
- The Rogers Center for Research & Training, Inc., Milwaukee, Wisconsin, United States